CLINICAL TRIAL: NCT04586023
Title: A Phase III Multicenter Randomized, Double-Blind, Double-Dummy, Parallel-Group Study to Evaluate the Efficacy and Safety of Fenebrutinib Compared With Teriflunomide in Adult Patients With Relapsing Multiple Sclerosis
Brief Title: Study to Evaluate the Efficacy and Safety of Fenebrutinib Compared With Teriflunomide in Relapsing Multiple Sclerosis (RMS)
Acronym: FENhance 2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GN42272; 2020-001168-28 (EudraCT Number); 2022-502618-95-00 (EU CTIS Number)
Record Dates: First submitted 2020-10-08; First posted 2020-10-14 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Relapsing Multiple Sclerosis
MeSH Terms: interventions — fenebrutinib; teriflunomide

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Sponsor will also be blinded.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fenebrutinib (Experimental): Participants will receive oral fenebrutinib with teriflunomide-matching placebo.
  Interventions: Drug: Fenebrutinib; Drug: Placebo
- Teriflunomide (Active Comparator): Participants will receive oral teriflunomide with fenebrutinib-matching placebo in a blinded fashion.
  Interventions: Drug: Teriflunomide; Drug: Placebo

INTERVENTIONS:
Drug: Fenebrutinib — Participants will receive fenebrutinib.
  Arms: Fenebrutinib
Drug: Teriflunomide — Participants will receive teriflunomide.
  Arms: Teriflunomide
Drug: Placebo — Participants will receive teriflunomide-matching placebo or fenebrutinib-matching placebo.

SUMMARY:
A study to evaluate the efficacy and safety of fenebrutinib on disability progression and relapse rate in adult participants with RMS. Eligible participants will be randomized 1:1 to either fenebrutinib or teriflunomide. At the end of the DBT phase (after disclosure of the DBT results), the Sponsor will determine whether or not to initiate the open-label extension phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* Expanded Disability Status Scale (EDSS) score of 0 - 5.5 at screening.
* A diagnosis of RMS in accordance with the revised 2017 McDonald Criteria.
* Ability to complete the 9-Hole Peg Test (9-HPT) for each hand in < 240 seconds.
* Ability to perform the Timed 25-Foot Walk Test (T25FWT) in <150 seconds.
* For female participants of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and refrain from donating eggs.
* For male participants: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and refrain from donating sperm.

OLE Inclusion Criteria:

* Completed the Double-Blind Treatment (DBT) phase of the study (remaining on study treatment; no other Disease-Modifying Therapy (DMT) administered) and who, in the opinion of the investigator, may benefit from treatment with fenebrutinib.
* Participants randomized to the teriflunomide treatment arm during the DBT phase must undergo the accelerated teriflunomide elimination procedure (ATEP) prior to the first administration of open-label fenebrutinib.
* For female participants of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and refrain from donating eggs.
* For male participants: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and refrain from donating sperm.

Exclusion Criteria:

* Disease duration of > 10 years from the onset of symptoms and an EDSS score at screening < 2.0.
* Female participants who are pregnant or breastfeeding, or intending to become pregnant.
* Male participants who intend to father a child during the study.
* A diagnosis of primary progressive MS (PPMS) or non-active secondary progressive MS (SPMS).
* Any known or suspected active infection at screening, including but not limited to a positive screening tests for Hepatitis B and C, an active or latent or inadequately treated infection with tuberculosis (TB), a confirmed or suspected progressive multifocal leukoencephalopathy (PML).
* History of cancer including hematologic malignancy and solid tumors within 10 years of screening.
* Known presence of other neurological disorders, that could interfere with the diagnosis of MS or assessments of efficacy or safety during the study and clinically significant cardiovascular, psychiatric, pulmonary, renal, hepatic, endocrine, metabolic or gastrointestinal disease.
* Rare hereditary problems of galactose intolerance, total lactase deficiency, or glucose-galactose malabsorption.
* Hypoproteinemia.
* Acute liver disease
* Chronic liver disease unless considered stable for > 6 months.
* Presence of cirrhosis (Child-Pugh Class A, B, or C) or Gilbert's Syndrome.
* Participants with significantly impaired bone marrow function or significant anemia, leukopenia, neutropenia or thrombocytopenia.
* Any concomitant disease that may require chronic treatment with systemic corticosteroids or immunosuppressants during the course of the study.
* History of alcohol or other drug abuse within 12 months prior to screening.
* History of or currently active primary or secondary (non-drug-related) immunodeficiency, including known history of human immunodeficiency virus (HIV) infection.
* Inability to complete an MRI scan.
* Adrenocorticotropic hormone or systemic corticosteroid therapy within 4 weeks prior to screening (inhaled and topical corticosteroids are allowed).
* Receipt of a live-attenuated vaccine within 6 weeks prior to randomization.
* Any previous treatment with immunomodulatory or immunosuppressive medication without an appropriate washout period.

OLE Exclusion Criteria:

* Chronic liver disease unless considered stable for > 6 months
* Acute liver disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 751 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2025-09-05 (Actual); Study Completion 2027-07-09 (Estimated)

PRIMARY OUTCOMES:
Annualized Relapse Rate (ARR) | Minimum of 96 weeks

SECONDARY OUTCOMES:
Time to Onset of Composite 12-week Confirmed Disability Progression (cCDP12) | Minimum of 96 weeks
Time to Onset of Composite 24-week Confirmed Disability Progression (cCDP24) | Minimum of 96 weeks
Time to Onset of 12-week Confirmed Disability Progression (CDP12) | Minimum of 96 weeks
Time to Onset of 24-week Confirmed Disability Progression (CDP24) | Minimum of 96 weeks
Total Number of T1 Gadolinium-enhancing (Gd+) Lesions, New and/or Enlarging T2-weighted Lesions as Detected by Magnetic Resonance Imaging (MRI) | Baseline, Weeks 12, 24, 48 and 96
Percentage Change in Total Brain Volume from Week 24 as Assessed by MRI | From Week 24 to Week 96
Change in Participant-Reported Physical Impacts of Multiple Sclerosis (MS) Measured by the Multiple Sclerosis, 29-Item [MSIS-29] Physical Scale | Baseline, Weeks 12, 24, 36, 48, 60, 72, 84 and 96
  The MSIS-29, version 2 is a 29-item patient-reported measure of the physical and psychological impacts of MS. Participants are asked to rate how much their functioning and well-being has been impacted over the past 14 days on a 4-point scale, from "Not at all" (1) to "Extremely" (4). The physical score is the sum of items 1-20, which is then transformed to a 0-100 scale. The psychological score is the sum of items 21-29, transformed to a 0-100 scale. Higher scores indicate a greater impact of MS.
Time to Onset of 12-week Confirmed 4-point Worsening in Symbol Digit Modality Test (SDMT) Score | Minimum of 96 weeks
  The SDMT is used for detecting the presence of cognitive impairment and changes in cognitive functioning over time and in response to treatment. The SDMT is brief, is easy to administer test, and involves a simple substitution task. Using a reference key, the examinee has 90 seconds to pair specific numbers with given geometric figures. Responses will be collected only orally, and administration time is approximately 5 minutes. The number of correct responses in 90 seconds will be considered the SDMT score. A decrease by 4 points on the SDMT score from baseline represents a clinically meaningful change in cognitive processing. The SDMT score ranges from 0 to 110. The higher the results, the better processing speed/working memory.
Change from Baseline to Week 48 in the Concentration of Blood Neurofilament Light chain (NfL) | Up to 48 weeks
Percentage of Participants with Adverse Events (AEs) | Up to 4.5 years
Plasma Concentrations of Fenebrutinib at Specified Timepoints | Up to 4.5 years
Time to Onset of Composite 12-week Confirmed Progression Independent of Relapse Activity (cPIRA12) | Minimum of 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (108):
- United States (13):
  - North Central Neurology Associates, Cullman, Alabama
  - Xenoscience, Phoenix, Arizona
  - Los Angeles Biomedical Research Institute at Harbor-UCLA, Torrance, California
  - KI Health Partners, LLC, Stamford, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - University of South Florida, Tampa, Florida
  - American Health Network Institute, LLC, Avon, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Neuro Institute of New England P.C., Foxborough, Massachusetts
  - University of Cincinnati, Cincinnati, Ohio
  - Hope Neurology, Knoxville, Tennessee
  - Integrated Neurology Services PLLC, Falls Church, Virginia
  - Medical College of Wisconsin, Inc., Milwaukee, Wisconsin
- Kepler Universitätskliniken GmbH - Med Campus III, Linz, Austria
- Brazil (12):
  - L2 Ip Instituto de Pesquisas Clinicas Ltda ME, Brasília, Federal District
  - Santa Casa de Misericordia, Belo Horizonte, Minas Gerais
  - Instituto de Neurologia de Curitiba, Curitiba, Paraná
  - IMV Pesquisa Neurológica, Porto Alegre, Rio Grande do Sul
  - Núcleo de Pesquisa do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Clinica Neurologica, Joinville, Santa Catarina
  - Praxis Pesquisa Médica, Santo André, São Paulo
  - CEMEC - Centro Multidisciplinar de Estudos Clínicos, São Bernardo do Campo, São Paulo
  - Centro de Pesquisas Clinicas, São Paulo, São Paulo
  - Hospital Santa Marcelina, São Paulo, São Paulo
  - Jordy Sinapse Medicina LTDA ME, São Paulo
- Bulgaria (2):
  - UMHAT Dr. Georgi Stranski, Pleven
  - MHATNP Sveti Naum EAD, Sofia
- Canada (5):
  - University of Alberta Hospital, Edmonton, Alberta
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - CIUSSS du Saguenay Lac-Saint-Jean, Chicoutimi Hospital, Chicoutimi, Quebec
  - MUCH - Montreal Neurological Institute & Hospital, Montreal, Quebec
  - CHU de Québec, Québec, Quebec
- Denmark (2):
  - Sydvestjysk Sygehus Esbjerg, Esbjerg
  - Hjerne- og nervesygdomme, Ambulatorium, Skleroseklinikken, Sønderborg
- France (4):
  - Hopital Gabriel Montpied CHU de Clermont-Ferrand, Clermont-Ferrand
  - Hôpital Pasteur, Nice
  - Hôpital Charles Nicolle, Rouen
  - CHU toulouse - Hôpital Purpan, Toulouse
- Greece (3):
  - Hospital Eginition, Athens
  - University General Hospital of Larisa, Larissa
  - AHEPA Univ. General Hospital of Thessaloniki, Thessaloniki
- Nucare, Guatemala City, Guatemala
- India (9):
  - Zydus Hospital, Ahmedabad, Gujarat
  - Seth G.S Medical College K.E.M Hospital, Mumbai, Maharashtra
  - Deenanath Mangeshkar Hospital & Research Centre, Pune, Maharashtra
  - Sahyadri Superspeciality Hospital, Pune, Maharashtra
  - Max Super Speciality Hospital, New Delhi, National Capital Territory of Delhi
  - Sir Gangaram Hospital, New Delhi, National Capital Territory of Delhi
  - Christian Medical College and Hospital, Ludhiana, Punjab
  - SRM Institute of Medical Sciences, Vadapalani, Tamil Nadu
  - Postgraduate Institute of Medical Education and Research, Chandigarh
- Italy (13):
  - Universita? G. D'Annunzio, Chieti, Abruzzo
  - Azienda Ospedaliero-Universitaria Consorziale Pol. di Bari, Bari, Apulia
  - A. O. U. Federico II, Napoli, Campania
  - Ospedale S.Camillo Forlanini, Rome, Lazio
  - Policlinico Universitario A. Gemelli, Rome, Lazio
  - NCL Institute Neuroscience, Rome, Lazio
  - Irccs A.O.U.San Martino Ist, Genoa, Liguria
  - Fond. Istituto Neurologico C.Besta, Milan, Lombardy
  - Ospedale Civile di Montichiari, Montichiari, Lombardy
  - IRCCS Istituto Neurologico C. Mondino?Dip. Neurologia Neuroriabilitazione S.S. Sclerosi Multipla, Pavia, Lombardy
  - IRCCS Istituto Neurologico Neuromed, Pozzilli, Molise
  - Ospedale Binaghi, Cagliari, Sardinia
  - AOU Policlinico Giaccone, Palermo, Sicily
- Mexico (5):
  - Mexico Centre for Clinical Research, Mexico City, Mexico CITY (federal District)
  - Clinstile S.A de C.V., Mexico City, Mexico CITY (federal District)
  - Grupo Médico Camino S.C., México, Mexico CITY (federal District)
  - Unidad de Investigación en Salud, Chihuahua City
  - Unidad de investigacion en salud (UIS), Mexico City
- Poland (15):
  - NZOZ Vitamed, Bydgoszcz
  - Neurocentrum Bydgoszcz sp. z o.o, Bydgoszcz
  - COPERNICUS Podmiot Leczniczy Sp. z o. o. Szpital im. M. Kopernika, Gdansk
  - RESMEDICA Spolka z o.o., Kielce
  - Centrum Neurologii Klinicznej, Krakow
  - Malopolskie Centrum Diagnostyczne MEDICAL Sp. z o. o., Krakow
  - Centrum Neurologii Krzysztof Selmaj, Lodz
  - Instytut Zdrowia Dr Boczarska-Jedynak Sp. z o.o. Sp. k., Oświęcim
  - Neurologiczny Niepubliczny ZOZ Centrum Leczenia SM Osrodek Bada? Klinicznych, Plewiska
  - MedPolonia, Poznan
  - NZOZ NEURO-KARD Ilkowski i Partnerzy Sp. Partn. Lek, Późna
  - Wojewódzki Szpital Specjalistyczny Nr 3, Rybnik
  - Klinika Neurologii I Wydzialu Lekarskiego WUM w Warszawie, Warsaw
  - Wro Medica, Wroc?aw
  - IBISMED Wielospecjalistyczne Centrum Medyczne, Zabrze
- Russia (7):
  - Krasnoyarsk State Medical Academy, Krasnoyarsk, Krasnoyarsk Krai
  - FSBHI Siberian Clinical Center of the Federal Medical and Biological Agency, Krasnoyarsk, Krasnoyarsk Krai
  - Federal center of brain research and neurotechnologies, Moskva, Moscow Oblast
  - Regional Clinical Hospital N.A. Semashko, Nizhny Novgorod, Niznij Novgorod
  - National Center of Social Significant Disease, Saint Petersburg, Sankt-Peterburg
  - Regional clinical hospital named after prof. S.V. Ochapovsky, Krasnodar
  - Nebbiolo Center for Clinical Trials, Tomsk
- South Korea (4):
  - Keimyung University Dongsan Medical Center, Daegu
  - National Cancer Center, Goyang-si
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
- Turkey (Türkiye) (11):
  - Gazi University Medical Faculty, Ankara
  - Baskent Universitesi Ankara Hastanesi, Çankaya
  - Bakirkoy State Mental Hospital, Istanbul
  - Sancaktepe Training and Research Hospital, Istanbul
  - Selcuk University Medical Faculty, Istanbul
  - Kocaeli University Hospital, Kocaeli
  - Ege Üniversitesi Tip Fakültesi, Lzmir
  - Mersin University Medical Faculty, Mersin
  - Ondokuz Mayis University School of Medicine, Samsun
  - Karadeniz Tecnical Uni. Med. Fac., Trabzon
  - Van Yuzuncu Yil University Hospital, Van
- Salford Royal NHS Foundation Trust, Salford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing